CLINICAL TRIAL: NCT06856590
Title: Impact of Zinc Supplementation and Transdermal Clobetasol in the Prophylaxis of Regorafenib-Induced Hand-Foot Skin Reaction: A Prospective Non-Randomized Study
Brief Title: ZINCLO-HAND: Zinc and Clobetasol for the Prevention of Regorafenib-Induced Hand-Foot Skin Reaction
Acronym: ZINCLO-HAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Orhun Akdoğan, MD, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AESH-EK-2025-042; Ankara Etlik City Hospital EC (Other: Republic of Türkiye Ministry of Health, Ankara Etlik City Hospital Ethics Committee)
Record Dates: First submitted 2025-02-21; First posted 2025-03-04 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-02

CONDITIONS: Hand-Foot Skin Reaction (HFSR)
Keywords: Regorafenib-Induced Skin Toxicity; Clobetasol; Zinc Supplementation; Metastatic Colorectal Cancer (mCRC); Gastrointestinal Stromal Tumor (GIST); Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Colorectal Neoplasms; Gastrointestinal Stromal Tumors; Carcinoma, Hepatocellular | interventions — Clobetasol

STUDY DESIGN:
Intervention Model Description: This study follows a parallel assignment model, where participants are assigned to one of three intervention groups based on the treating physician's decision. Each group receives a different preventive approach for regorafenib-induced hand-foot skin reaction (HFSR):
  1. Oral zinc supplementation + transdermal clobetasol cream
  2. Transdermal clobetasol cream alone
  3. Oral zinc supplementation alone
  Participants will remain in their assigned groups throughout the study period, and no crossover between groups will occur. The study aims to compare the efficacy of these interventions in preventing and reducing the severity of HFSR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Zinc + Clobetasol Group (Experimental): Participants in this group will receive oral zinc supplementation (78 mg zinc gluconate twice daily) combined with topical clobetasol propionate 0.05% cream, applied twice daily to the palms and soles for 8 weeks. This group aims to evaluate the combined efficacy of zinc and clobetasol in preventing regorafenib-induced hand-foot skin reaction (HFSR).
  Interventions: Dietary Supplement: Zinc Supplementation; Drug: Clobetasol Propionate 0.05% Cream
- Clobetasol Alone Group (Experimental): Participants in this group will receive topical clobetasol propionate 0.05% cream, applied twice daily to the palms and soles for 8 weeks. This group aims to assess the efficacy of clobetasol alone in preventing regorafenib-induced HFSR.
  Interventions: Drug: Clobetasol Propionate 0.05% Cream
- Zinc Alone (Experimental): Participants in this group will receive oral zinc supplementation (78 mg zinc gluconate twice daily) for 8 weeks. This group aims to determine the role of zinc alone in reducing the severity of regorafenib-induced HFSR.
  Interventions: Dietary Supplement: Zinc Supplementation

INTERVENTIONS:
Dietary Supplement: Zinc Supplementation — Participants assigned to zinc-containing arms will receive oral zinc gluconate supplementation (78 mg twice daily) for 8 weeks. This intervention aims to evaluate the effect of zinc in preventing and reducing the severity of regorafenib-induced hand-foot skin reaction (HFSR).
  Arms: Zinc + Clobetasol Group; Zinc Alone
Drug: Clobetasol Propionate 0.05% Cream — Participants assigned to clobetasol-containing arms will receive topical clobetasol propionate 0.05% cream, applied twice daily to the palms and soles for 8 weeks. This intervention aims to assess the efficacy of clobetasol in preventing regorafenib-induced HFSR.
  Arms: Clobetasol Alone Group; Zinc + Clobetasol Group

SUMMARY:
This study aims to evaluate whether a combination of oral zinc supplementation and transdermal clobetasol cream is effective in preventing and reducing the severity of hand-foot skin reaction (HFSR) induced by regorafenib treatment.

HFSR is one of the most common adverse effects of regorafenib, affecting more than 50% of patients, with 10-15% experiencing severe Grade 3 toxicity. Clobetasol, a high-potency corticosteroid, has been shown to significantly reduce the severity of HFSR when used preemptively rather than reactively. Additionally, recent clinical trials indicate that oral zinc supplementation may further reduce the incidence of Grade ≥2 HFSR.

This prospective, non-randomized interventional study will compare three treatment groups:

Oral zinc supplementation + transdermal clobetasol cream Transdermal clobetasol cream alone Oral zinc supplementation alone The study will assess the effectiveness of these treatments using CTCAE grading, the Hand-Foot Syndrome Scale-14, and quality of life measures (FACT-G, fatigue, and anxiety/depression scales). Additionally, the study will evaluate the impact of HFSR on treatment adherence, regorafenib dose modifications, and overall survival.

The study will enroll approximately 120 patients across multiple centers in Türkiye.

DETAILED DESCRIPTION:
Background and Rationale Hand-foot skin reaction (HFSR) is a common dose-limiting toxicity associated with regorafenib treatment, occurring in more than 50% of patients and leading to treatment modifications in up to 15% of cases. Despite its clinical significance, no standardized prophylactic strategy exists.

High-potency topical corticosteroids, such as clobetasol propionate 0.05%, have demonstrated efficacy in reducing HFSR severity, particularly when used preemptively. Additionally, recent studies suggest that oral zinc supplementation may contribute to maintaining skin integrity and reducing inflammatory responses, thereby mitigating HFSR severity. However, the comparative efficacy of these interventions and their potential synergistic effect have not been well established.

Study Objectives This study aims to evaluate whether oral zinc supplementation and/or transdermal clobetasol cream effectively prevent and reduce the severity of regorafenib-induced HFSR, thereby improving treatment adherence and patient quality of life.

Study Design

This is a prospective, non-randomized, interventional study involving approximately 120 patients receiving regorafenib at multiple oncology centers in Türkiye. Participants will be assigned to one of three intervention arms based on their treating physician's discretion:

Oral zinc supplementation + transdermal clobetasol cream Transdermal clobetasol cream alone Oral zinc supplementation alone Interventions Oral Zinc Supplementation: 78 mg zinc gluconate, administered twice daily for 8 weeks.

Transdermal Clobetasol Cream: Clobetasol propionate 0.05%, applied twice daily to the palms and soles for 8 weeks.

Assessment & Follow-up HFSR severity and incidence will be evaluated using CTCAE v5.0 criteria. Patient-reported outcomes will be assessed via Hand-Foot Syndrome Scale-14 (HFS-14) and FACT-G quality of life questionnaire.

Regorafenib adherence (dose modifications, treatment discontinuations) will be monitored.

Survival analysis (PFS and OS) will be conducted at 6 months. By comparing these prophylactic strategies, this study seeks to identify the most effective approach to minimize HFSR burden in patients undergoing regorafenib therapy, potentially influencing future clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed solid tumor for which regorafenib is an approved treatment (e.g., metastatic colorectal cancer, gastrointestinal stromal tumor, hepatocellular carcinoma, glioblastoma, or others)
* Initiating regorafenib treatment for the first time
* ECOG performance status of 0-2
* Baseline hand-foot skin reaction (HFSR) of Grade 0 (no prior HFSR symptoms) according to CTCAE v5.0
* Adequate organ function, including:

AST/ALT ≤ 3× upper limit of normal (ULN) Creatinine clearance > 50 mL/min Hemoglobin ≥ 9 g/dL Platelet count ≥ 75,000/mm³

* Able to tolerate oral zinc supplementation and/or topical corticosteroids
* Willing to participate and provide informed consent

Exclusion Criteria:

* Pre-existing dermatologic conditions affecting the hands or feet (e.g., psoriasis, eczema, active infections)
* Prior Grade ≥1 HFSR from any VEGFR-TKI therapy
* Allergy or known hypersensitivity to zinc, clobetasol, or other study components

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-07 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Hand-Foot Skin Reaction (HFSR) at Week 8 | 8 weeks
  The incidence and severity of hand-foot skin reaction (HFSR) will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The proportion of patients experiencing Grade ≥2 HFSR will be compared between the intervention groups to evaluate the efficacy of zinc supplementation and/or clobetasol in preventing HFSR.

SECONDARY OUTCOMES:
Duration of Hand-Foot Skin Reaction (HFSR) | 8 weeks
  The time from the onset of Grade ≥2 HFSR to its resolution (return to Grade 1 or lower) will be measured in each intervention group. The effectiveness of zinc supplementation and/or clobetasol in shortening HFSR duration will be evaluated.
Regorafenib Dose Modifications Due to HFSR | 8 weeks
  The percentage of participants requiring dose reduction, dose delay, or treatment discontinuation due to HFSR will be recorded. The impact of prophylactic zinc supplementation and/or clobetasol on maintaining regorafenib treatment adherence will be assessed.
Quality of Life (FACT-G Score Change) | Baseline and 8 weeks
  Changes in quality of life (QoL) will be assessed using the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire. QoL scores at baseline and at Week 8 will be compared among the intervention groups. The FACT-G total score ranges from 0 to 108, with higher scores indicating better quality of life.
Progression-Free Survival (PFS) in Patients with and without Severe HFSR | Up to 6 months
  The time from the start of regorafenib treatment to disease progression or death from any cause, whichever occurs first.
Overall Survival (OS) in Patients with and without Severe HFSR | 6 months
  The time from the start of regorafenib treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ozan Yazıcı, Prof., Study Chair — Gazi University
Locations (13):
- Turkey (Türkiye) (13):
  - Necmettin Erbakan University Meram Faculty of Medicine Hospital, Konya, Meram
  - Bursa Uludağ University Hospital, Bursa, Nilüfer
  - Karadeniz Technical University Hospital, Trabzon, Ortahisar
  - Sakarya University Hospital, Sakarya, Serdivan
  - Ankara Etlik City Hospital, Ankara, Yenimahalle
  - Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara, Yenimahalle
  - Gazi University, Ankara, Yenimahalle
  - Afyonkarahisar University of Health Sciences Hospital, Afyonkarahisar
  - Ankara University Faculty of Medicine Hospital, Ankara
  - Hacettepe University Faculty of Medicine Hospital, Ankara
  - Dicle University Hospital, Diyarbakır
  - Tekirdağ Namık Kemal University Hospital, Tekirdağ
  - Van Yüzüncü Yıl University Dursun Odabaş Hospital, Van

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy regulations and institutional policies. Data access is restricted to the study team and authorized personnel to ensure compliance with ethical guidelines and patient confidentiality